CLINICAL TRIAL: NCT00321737
Title: A Phase 3 Study to Evaluate the Safety and Efficacy of TAK-390MR (30 mg QD and 60 mg QD) Compared to Placebo in Maintenance of Healing in Subjects With Healed Erosive Esophagitis.
Brief Title: Efficacy and Safety of Dexlansoprazole MR Compared to Placebo on Maintaining Healing in Subjects With Healed Erosive Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T-EE05-135; 2006-000419-90 (EudraCT Number); U1111-1113-9433 (Registry Identifier: WHO)
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Results first posted 2009-08-28 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Esophagitis, Reflux; Esophagitis, Peptic
Keywords: Erosive Esophagitis
MeSH Terms: conditions — Esophagitis, Peptic | interventions — Dexlansoprazole; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexlansoprazole MR 30 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole MR
- Dexlansoprazole MR 60 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole MR
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexlansoprazole MR — Dexlansoprazole MR 30 mg, capsules, orally, once daily for up to six months.
  Other Names: TAK-390MR; Kapidex; Dexilant
  Arms: Dexlansoprazole MR 30 mg QD
Drug: Dexlansoprazole MR — Dexlansoprazole MR 60 mg, orally, once daily for up to six months.
  Other Names: TAK-390MR; Kapidex; Dexilant
  Arms: Dexlansoprazole MR 60 mg QD
Drug: Placebo — Dexlansoprazole placebo-matching capsules, orally, once daily for up to six months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the ability of once-daily (QD) treatment with dexlansoprazole modified release (MR) 30 mg and 60 mg or placebo in maintaining healing of erosive esophagitis (EE).

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, multicenter, placebo-controlled, 6 month maintenance study. The study is designed to compare the efficacy and safety of daily dexlansoprazole MR (30 mg and 60 mg) with that of placebo, in maintaining healing of EE.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have successfully completed the Phase 3 Study T-EE04-084 (NCT00251693) or T-EE04-085 (NCT00251719); and have healed esophageal erosions proven by endoscopy. Complete healing was assessed for change in LA Esophagitis Classification grades A, B, C, or D to healed (defined as anything less than the criterion for Grade A). The subject was counted as healed if endoscopy findings did not meet the Grade A criterion.

Exclusion Criteria:

* Use of prescription or nonprescription proton pump inhibitors (PPIs), histamine (H2) receptor antagonists, sucralfate, misoprostol, or prokinetics throughout the study.
* Use of antacids (except for study supplied) throughout the study.
* Use of drugs with significant anticholinergic effects such as tricyclics who cannot stay on a stable dose throughout the study.
* Chronic (>12 doses per month) use of nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclo-oxygenase-2 (COX-2) inhibitors.
* Need for continuous anticoagulant therapy.
* Evidence of uncontrolled systemic disease.
* Subjects who have participated in either maintenance study (T-EE04-086 [NCT00255164] or T-EE04-087 [NCT00255151]).
* Subjects who, in the opinion of the investigator, is unable to comply with the requirements of the study or is unsuitable for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Takeda
Locations (98):
- United States (80):
  - Huntsville, Alabama
  - Tuscon, Arizona
  - Anaheim, California
  - Azusa, California
  - Carmichael, California
  - Chula Vista, California
  - Cypress, California
  - Fresno, California
  - Garden Grove, California
  - Harrisburg, California
  - Irvine, California
  - Lancaster, California
  - Mission Hills, California
  - Oakland, California
  - Orange, California
  - Pasadena, California
  - San Diego, California
  - San Luis Obispo, California
  - Boulder, Colorado
  - Colorado Springs, Colorado
  - Wheat Ridge, Colorado
  - Boynton Beach, Florida
  - Jupiter, Florida
  - Miami, Florida
  - New Smyma Beach, Florida
  - Ocala, Florida
  - St. Petersburg, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Boise, Idaho
  - Moline, Illinois
  - Oak Forrest, Illinois
  - Rockford, Illinois
  - Clive, Iowa
  - Lexington, Kentucky
  - Baton Rouge, Louisiana
  - Metairie, Louisiana
  - Chevy Chase, Maryland
  - Hollywood, Maryland
  - Lutherville, Maryland
  - Prince Federick, Maryland
  - Chaska, Minnesota
  - Jackson, Mississippi
  - Jefferson City, Missouri
  - Washington, Missouri
  - Egg Harbor, New Jersey
  - Albuquerque, New Mexico
  - Binghamton, New York
  - Rochester, New York
  - Greensboro, North Carolina
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Bismarck, North Dakota
  - Dayton, Ohio
  - Mogadore, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Duncansville, Pennsylvania
  - Lansdale, Pennsylvania
  - Anderson, South Carolina
  - Mt. Pleasant, South Carolina
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Jackson, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Ogden, Utah
  - Charlottesville, Virginia
  - Chesapeake, Virginia
  - Spokane, Washington
  - Tacoma, Washington
  - Milwaukee, Wisconsin
  - Monroe, Wisconsin
- Kippa-Ring, Australia
- Canada (6):
  - St. John's, Newfoundland and Labrador
  - Newmarket, Ontario
  - Richmond Hill, Ontario
  - Toronto, Ontario
  - Longueuil, Quebec
  - Regina, Saskatchewan
- Hradec Králové, Czechia
- Tallinn, Estonia
- Latvia (2):
  - Riga
  - Valmiera
- Lithuania (3):
  - Kaunas
  - Panevezys
  - Vilnius
- Slovakia (4):
  - Bratislava
  - Nitra
  - Prešov
  - Sučany

REFERENCES:
- [Result] Metz DC, Howden CW, Perez MC, Larsen L, O'Neil J, Atkinson SN. Clinical trial: dexlansoprazole MR, a proton pump inhibitor with dual delayed-release technology, effectively controls symptoms and prevents relapse in patients with healed erosive oesophagitis. Aliment Pharmacol Ther. 2009 Apr 1;29(7):742-54. doi: 10.1111/j.1365-2036.2009.03954.x. Epub 2009 Feb 7. PMID 19210298
- [Result] Peura DA, Metz DC, Dabholkar AH, Paris MM, Yu P, Atkinson SN. Safety profile of dexlansoprazole MR, a proton pump inhibitor with a novel dual delayed release formulation: global clinical trial experience. Aliment Pharmacol Ther. 2009 Nov 15;30(10):1010-21. doi: 10.1111/j.1365-2036.2009.04137.x. Epub 2009 Sep 4. PMID 19735233
- [Result] Wyrwich KW, Mody R, Larsen LM, Lee M, Harnam N, Revicki DA. Validation of the PAGI-SYM and PAGI-QOL among healing and maintenance of erosive esophagitis clinical trial participants. Qual Life Res. 2010 May;19(4):551-64. doi: 10.1007/s11136-010-9620-x. Epub 2010 Feb 27. PMID 20195905
- [Result] Friedlander EA, Pallentino J, Miller SK, VanBeuge SS. The evolution of proton pump inhibitors for the treatment of gastroesophageal reflux disease. J Am Acad Nurse Pract. 2010 Dec;22(12):674-83. doi: 10.1111/j.1745-7599.2010.00578.x. Epub 2010 Nov 24. PMID 21129076
- See also: For the Dexilant package insert refer to this link — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=9efb34b3-fb69-4190-a2be-a90b8cb94e25&filetypecode=DEXILANTPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at a total of 94 sites: 75 sites in the United States and 19 sites in Australia, Canada, the Czech Republic, Estonia, India, Latvia, Lithuania, Poland, and the Slovak Republic (date of first dose: 19 May 2006; date of last procedure: 21 May 2007).
Pre-assignment Details: Subjects had to have endoscopically proven healed erosive esophagitis (EE) after 4 to 8 weeks of treatment with lansoprazole 30 mg once-daily (QD), dexlansoprazole modified release (MR) 60 mg QD, or dexlansoprazole MR 90 mg QD in the EE healing studies, T-EE04-084 (NCT00251693) and T-EE04-085 (NCT00251719).
Groups:
- Placebo QD: Placebo capsules, orally, once daily for up to 6 months.
- Dexlansoprazole MR 30 mg QD: Dexlansoprazole MR 30 mg, capsules, orally, once daily for up to 6 months.
- Dexlansoprazole MR 60 mg QD: Dexlansoprazole MR 60 mg, capsules, orally, once daily for up to 6 months.
Period: Overall Study
Arm/Group | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Started | 147 | 140 | 158
Completed | 25 | 92 | 104
Not Completed | 122 | 48 | 54
Not completed — Relapse of Erosive Esophagitis | 76 | 25 | 19
Not completed — Adverse Event | 11 | 3 | 6
Not completed — Lost to Follow-up | 5 | 5 | 6
Not completed — Withdrawal by Subject | 19 | 12 | 17
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Unmet Inclusion/Exclusion Criteria | 1 | 0 | 0
Not completed — Possible Barrett's Esophagus | 2 | 1 | 1
Not completed — Therapeutic Failure | 6 | 0 | 2
Not completed — Pregnancy | 0 | 2 | 0
Not completed — Noncompliance | 2 | 0 | 0
Not completed — Subject Request/ Subject Unavailable | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD | Total
Number analyzed (Participants) | 147 | 140 | 158 | 445
Age Continuous [Mean (Standard Deviation); unit: years] | 49.5 (12.94) | 47.1 (13.15) | 47.9 (11.72) | 48.2 (12.60)
Age, Customized [Number; unit: participants]
  <45 years | 50 | 54 | 58 | 162
  45 - <65 years | 83 | 75 | 89 | 247
  ≥65 years | 14 | 11 | 11 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 71 | 84 | 230
  Male | 72 | 69 | 74 | 215
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 4 | 4
  Asian | 3 | 3 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 4 | 6 | 11 | 21
  White | 138 | 127 | 135 | 400
  More than one race | 1 | 4 | 2 | 7
  Unknown or Not Reported | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 21 | 19 | 60
  Not Hispanic or Latino | 127 | 119 | 139 | 385
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline Los Angeles (LA) Classification Grade for Erosive Esophagitis (EE) [Number; unit: participants] — Baseline values from Studies T-EE04-084 (NCT00251693) and T-EE04-085 (NCT00251719), with severity of EE increasing from Grade A to Grade D.
  participants
    A: ≥1 mucosal break <5 mm | 51 | 53 | 56 | 160
    B: ≥1 mucosal break ≥5 mm | 57 | 46 | 57 | 160
    C: ≥1 mucosal break <75% of circumference | 34 | 31 | 39 | 104
    D: ≥1 mucosal break ≥75% of circumference | 5 | 10 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Maintained Complete Healing of Erosive Esophagitis as Assessed by Endoscopy - Crude Rate Analysis.
Description: Crude rates analyzed maintenance of healed EE from baseline of this study and considered prematurely discontinued subjects as relapsed.
Time Frame: 6 months
Population: The crude rate analysis was performed on intent-to-treat (ITT) subjects (subjects from Studies T-EE04-084 or T-EE04-085 with endoscopically proven healed EE who received at least 1 dose of study drug in this study and did not have a gap of >7 days between the EE healing studies and this study) with at least one endoscopy in this maintenance study.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 119 | 125 | 143
Percentage of Subjects | 14.3 [8.4 to 22.2] | 66.4 [58.3 to 73.9] | 66.4 [55.9 to 72.4]
Statistical Analysis 1: Comparison: Placebo QD vs Dexlansoprazole MR 30 mg QD; Test type: Superiority or Other; p < 0.00001, Fisher Exact — Hochberg's method was used to ensure that the overall 0.0025 level of significance was maintained for the pairwise comparisons between each dexlansoprazole MR dose and placebo
Statistical Analysis 2: Comparison: Placebo QD vs Dexlansoprazole MR 60 mg QD; Test type: Superiority or Other; p < 0.00001, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 30 mg QD vs Dexlansoprazole MR 60 mg QD; Test type: Superiority or Other; p > 0.99999, Fisher Exact — Statistical significance was determined at the 0.0025 level without adjustment for multiple comparisons

2. Secondary Outcome: Percentage of Days Without Daytime or Nighttime Heartburn as Assessed by Daily Diary-Median.
Description: The percentage was calculated as the days that were heartburn-free out of the total number of days for which either a daytime or nighttime result was reported.
Time Frame: 6 months
Population: The analysis of 24-hour heartburn-free days was performed on ITT subjects with at least one daytime or nighttime heartburn Yes/No question answered during treatment.
Measure: Median (Inter-Quartile Range); unit: Percentage of Days
Arm/Group | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 141 | 132 | 147
Percentage of Days | 28.6 (32.0) [5.9 to 61.8] | 96.1 (26.5) [80.7 to 100.0] | 90.9 (28.3) [66.7 to 99.4]
Statistical Analysis 1: Comparison: Placebo QD vs Dexlansoprazole MR 30 mg QD; Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney) — The 0.0025 level of significance for this secondary endpoint was controlled using Hochberg's method for comparison of each dexlansoprazole MR dose to placebo
Statistical Analysis 2: Comparison: Placebo QD vs Dexlansoprazole MR 60 mg QD; Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 30 mg QD vs Dexlansoprazole MR 60 mg QD; Test type: Superiority or Other; p = 0.06730, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.0025 level without adjustment for multiple comparisons

3. Secondary Outcome: Percentage of Days Without Daytime or Nighttime Heartburn as Assessed by Daily Diary-Mean.
Description: The percentage was calculated as the days that were heartburn-free out of the total number of days for which either a daytime or nighttime result was marked.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of Days
Arm/Group | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 141 | 132 | 147
Percentage of Days | 36.0 (32.0) | 83.3 (26.5) | 78.4 (28.3)

4. Primary Outcome: Percentage of Subjects Who Maintained Complete Healing of Erosive Esophagitis as Assessed by Endoscopy - Life Table Method
Description: Percentage of subjects who maintained complete healing of erosive esophagitis as assessed by endoscopy. In the life table method, subjects without post-baseline endoscopy were included as censored; subjects who did not have a recurrence of EE and did not complete the study were also considered censored.
Time Frame: 6 months
Population: Life table method for the maintenance rate of healed EE was performed on ITT subjects and included subjects without post-baseline endoscopy as censored.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 145 | 137 | 153
Percentage of Subjects | 27.2 | 74.9 | 82.5
Statistical Analysis 1: Comparison: Placebo QD vs Dexlansoprazole MR 30 mg QD; Test type: Superiority or Other; p < 0.00001, Log Rank — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Dexlansoprazole MR 60 mg QD; Test type: Superiority or Other; p < 0.00001, Log Rank — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 30 mg QD vs Dexlansoprazole MR 60 mg QD; Test type: Superiority or Other; p = 0.13932, Log Rank — Statistical significance was determined at the 0.0025 level without adjustment for multiple comparisons

5. Secondary Outcome: Percentage of Days Without Nighttime Heartburn as Assessed by Daily Diary-Median.
Description: The percentage was calculated as the nights that were heartburn-free out of the total number of days for which a nighttime result was marked.
Time Frame: 6 months
Population: The analysis was performed on ITT subjects with at least one nighttime heartburn Yes/No question answered during treatment.
Measure: Median (Inter-Quartile Range); unit: Percentage of Days
Arm/Group | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 140 | 132 | 147
Percentage of Days | 71.7 (36.6) [19.5 to 92.2] | 98.9 (22.3) [90.9 to 100.0] | 96.2 (23.1) [80.0 to 100.0]
Statistical Analysis 1: Comparison: Placebo QD vs Dexlansoprazole MR 30 mg QD; Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney) — The 0.0025 level of significance for this secondary endpoint was controlled using Hochberg's method for comparison of each dose to placebo
Statistical Analysis 2: Comparison: Placebo QD vs Dexlansoprazole MR 60 mg QD; Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 30 mg QD vs Dexlansoprazole MR 60 mg QD; Test type: Superiority or Other; p = 0.11257, Wilcoxon (Mann-Whitney) — Statistical significance was determined at the 0.0025 level without adjustment for multiple comparisons

6. Secondary Outcome: Percentage of Days Without Nighttime Heartburn as Assessed by Daily Diary-Mean.
Description: as for outcome 5
Time Frame: 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of Days
Arm/Group | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 140 | 132 | 147
Percentage of Days | 57.7 (36.6) | 89.3 (22.3) | 86.0 (23.1)

ADVERSE EVENTS:
Arm/Group | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Serious Adverse Events (participants affected / at risk) | 1 | 2 | 6
Other Adverse Events (participants affected / at risk) | 11 | 26 | 35
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Implant and Catheter Site Reactions (General disorders) | 0/147 | 0/140 | 1/158
Pain and Discomfort Not Elsewhere Classified (NEC) (General disorders) | 0/147 | 0/140 | 1/158
Cholecystitis and Cholelithiasis (Hepatobiliary disorders) | 0/147 | 0/140 | 1/158
Bacterial Infections NEC (Infections and infestations) | 0/147 | 0/140 | 1/158
Viral Infections NEC (Infections and infestations) | 0/147 | 0/140 | 1/158
Limb Injuries NEC (Including [Incl] Traumatic Amputation) (Injury, poisoning and procedural complications) | 0/147 | 0/140 | 1/158
Non-Site Specific Injuries NEC (Injury, poisoning and procedural complications) | 0/147 | 0/140 | 1/158
Prostatic Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/147 | 1/140 | 0/158
Cerebrovascular Venous and Sinus Thrombosis (Nervous system disorders) | 0/147 | 0/140 | 1/158
Migraine Headaches (Nervous system disorders) | 0/147 | 0/140 | 1/158
Abortions Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/147 | 1/140 | 0/158
Ovarian And Fallopian Tube Cysts and Neoplasms (Reproductive system and breast disorders) | 0/147 | 0/140 | 1/158
Uterine Disorders NEC (Reproductive system and breast disorders) | 0/147 | 0/140 | 1/158
Bronchospasm and Obstruction (Respiratory, thoracic and mediastinal disorders) | 0/147 | 0/140 | 1/158
Peripheral Embolism and Thrombosis (Vascular disorders) | 0/147 | 0/140 | 1/158
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Diarrhoea (Excluding [Excl] Infective) (Gastrointestinal disorders) | 1/147 | 5/140 | 8/158
Gastritis (Excl Infective) (Gastrointestinal disorders) | 7/147 | 2/140 | 8/158
Upper Respiratory Tract Infections (Infections and infestations) | 1/147 | 14/140 | 17/158
Joint Related Signs and Symptoms (Musculoskeletal and connective tissue disorders) | 1/147 | 7/140 | 0/158
Musculoskeletal and Connective Tissue Signs and Symptoms NEC (Musculoskeletal and connective tissue disorders) | 2/147 | 3/140 | 8/158

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.